CLINICAL TRIAL: NCT06978309
Title: Exploring the Difference in EMG Response of Forearm and Sternocleidomastoid Muscles When Comparing Laparoscopic Surgery (LS) and Robot Assisted Laparoscopic Surgery (RALS).
Brief Title: EMG Response in Forearm and Neck Muscles When Comparing Surgical Techniques.
Status: Completed | Type: Observational
Sponsor: Lancaster University (Other)
Responsible Party: Principal Investigator, Matthew Davitt, Principal Investigator, Lancaster University
Other Study IDs: FHM-2025-4948-IRAS-2
Record Dates: First submitted 2025-04-23; First posted 2025-05-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Surgical Fatigue
Keywords: fatigue; Laparoscopic; Surgeon wellbeing; Robotic surgery; EMG
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robot-Assisted Laparoscopic Surgery: Surgeons performing robot assisted laparoscopic surgery.
  Interventions: Other: No Interventions
- Laparoscopic Surgery: Surgeons performing manual laparoscopic surgery.
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — Observational study.

SUMMARY:
Surgeons are performing an increasing number of minimal access procedures because these offer certain advantages including improved recovery times. However, this also results in surgeons operating for longer periods which inevitably increases the already known prevalence of work-related Musculoskeletal (MSK) injuries amongst surgeons. Work-related MSK disorders account for 26 - 47.5% of illnesses and injuries due to overexertion and repetitive use, in professionals with ergonomically challenging jobs. Robotic-assisted laparoscopic surgery (RALS) is a modern technology that could help mitigate these MSK problems and thereby improve patient care. In comparison to standard laparoscopic surgery (LS), RALS offers steadier wrist movements with a reduced fulcrum effect, thus benefiting the patient.

No study has compared the demands of RALS vs. LS on musculoskeletal fatigue (and subsequent injury risk). The investigators need to determine whether a career using RALS is associated with better musculoskeletal health of surgeons than standard LS when performing complex minimally invasive procedures.

The study will recruit Surgeons who perform prostate and bowel surgical procedures who have experience using RALS and/or LS. Surgeons will complete a series of validated questionnaires before and after each surgery to subjectively determine musculoskeletal strain/pain and will have body composition quantified.

They will be fitted with EMG (to measure muscle fatigue) whilst performing real-life surgery. Analysis of data gathered will be used to show what the short- and long- term musculoskeletal demands are and in turn determine if these are associated with changes in motor control.

The researcher's postulated hypothesis is that RALS should have less musculoskeletal effects both short and long term on surgeons, therefore, highlighting the fact that the implementation of RALS should be less controversial, because in the long run, the most expensive objects in the operating room are the personnel.

ELIGIBILITY:
Inclusion Criteria

* Either a laparoscopic or robot-assisted laparoscopic surgeon.
* Good musculoskeletal health.
* Adult.

Exclusion Criteria:

* Procedures with major complications (above 50% more time than the average for that surgery).
* Significant co- morbidities that could affect the results of the study. Significant symptoms of musculoskeletal disorder.
* Anything the investigator feels will affect the study's measurements of safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, adult laparoscopic and robot- assisted laparoscopic surgeons.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Acute muscle activation- percentage of forearm maximal voluntary contraction (%) assessed using EMG frequency. | Intraoperative
  This outcome measures the immediate impact of RALS and LS on the surgeon's forearm muscles during a single surgical procedure. It will be quantified by assessing the change in electromyography (EMG) frequency and amplitude recorded during clinically important surgical tasks within the surgeons' first surgery of the day. The contributing measures to this primary measure are the maximal voluntary contraction that will be assessed just before the surgery begins, and the average frequency of muscle activation (mV) over the 2 minute data collection period. Muscle activation for RALS and LS will be compared using this measure.

SECONDARY OUTCOMES:
Surgeon musculoskeletal health over the last 12 months (Standardized Nordic Questionnaire) | Preoperative
  This questionnaire assesses musculoskeletal symptoms experienced by the surgeons within the last 12 months. It helps to understand the prevalence and location of pain and discomfort before they participate in the study. This questionnaire primarily yields categorical data. For each of the nine body regions (neck, shoulders, upper back, elbows, low back, wrists/hands, hips/thighs, knees, ankles/feet), it asks about trouble (ache, pain, discomfort) in the past 12 months and in the past 7 days. It also asks if the trouble prevented normal work (at home or away from home).
Surgeon physical activity participation status (International Physical Activity Questionnaire | Preoperative
  The frequency, duration, and intensity of different types of physical activities (vigorous, moderate, walking, and sitting) undertaken by the surgeons. It aims to quantify their overall physical activity level. Can be reported as continuous scores (Metabolic Equivalent of Task - minutes per week, or MET-min/week) calculated by multiplying duration, frequency, and standard MET intensity values for each activity type. It can also be categorized into low, moderate, and high physical activity levels based on specific criteria related to frequency, duration, and total MET-min/week.
Surgeon well-being and quality of life (SF36 Health and Wellbeing Questionnaire) | Preoperative
  This assesses the surgeon's health-related quality of life across eight dimensions: Physical Functioning, Role Limitations due to Physical Health Problems, Bodily Pain, General Health Perceptions, Vitality (energy/fatigue), Social Functioning, Role Limitations due to Emotional Problems,1 and Mental Health (emotional well-being). This yields eight scaled scores ranging from 0 to 100, with higher scores indicating better health status in each dimension. Scoring involves recoding items, summing within scales, and then transforming to the standardized range using specific algorithms. Summary scores (PCS and MCS) can also be calculated.
Maximal Voluntary Contraction measured using EMG (mV) | Intraoperative
  This will take place with the surgeon producing the a maximal contraction for both their forearm muscles and neck muscles in to create a baseline of comparison to calculate the percentage of maximal contraction that the surgeons experience during surgery.
Acute muscle activation- percentage of sternocleidomastoid maximal voluntary contraction (%) assesed using EMG frequency. | Intraoperative
  This outcome measures the immediate impact of RALS and LS on the surgeon's sternocleidomastoid muscles during a single surgical procedure. It will be quantified by assessing the change in electromyography (EMG) frequency and amplitude recorded during clinically important surgical tasks within the surgeons' first surgery of the day. The contributing measures to this primary measure are the maximal voluntary contraction that will be assessed just before the surgery begins, and the average frequency of muscle activation (mV) over the 2 minute data collection period. Muscle activation for RALS and LS will be compared using this measure.
Average sternocleidomastoid and forearm muscle EMG amplitude (mV) | Intraoperative
  This will be measured using EMG at clinically significant points in the surgery. This will allow for the researchers to assess the muscular demand and the amplitude and frequency of the EMG signal are the direct measures used to quantify this primary variable. Lower amplitude means a greater muscular demand.
Average sternocleidomastoid and forearm muscle EMG frequency (Hz). | Intraoperative
  This will be measured using EMG at clinically significant points in the surgery. This will allow for the researchers to assess the muscular demand and the amplitude and frequency of the EMG signal are the direct measures used to quantify this primary variable. Higher frequency means greater muscular demand.
Surgeon musculoskeletal health over the last 12 months (Standardized Nordic Questionnaire) | Any time between enrolment in the study and the date of the surgical procedure that the data collection will take place.
  This questionnaire assesses musculoskeletal symptoms experienced by the surgeons within the last 12 months. It helps to understand the prevalence and location of pain and discomfort before they participate in the study. This questionnaire primarily yields categorical data. For each of the nine body regions (neck, shoulders, upper back, elbows, low back, wrists/hands, hips/thighs, knees, ankles/feet), it asks about trouble (ache, pain, discomfort) in the past 12 months and in the past 7 days. It also asks if the trouble prevented normal work (at home or away from home).

CONTACTS AND LOCATIONS:
Locations (1):
- Blackburn Royal Teaching Hospital, Blackburn, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Only IPD in the published results will potentially be included.

DOCUMENTS (1):
  • Study Protocol (2025-09-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT06978309/Prot_000.pdf